CLINICAL TRIAL: NCT00238888
Title: Randomised Controlled Trial of a Multi-faceted Community-based Intervention to Improve Pediatric Morbidity: a PRIISME Project (Program to Integrate Information Service and Manage Education)
Brief Title: Randomised Controlled Trial of a Multi-faceted Community-based Intervention to Improve Asthma in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Francine Ducharme, Francine Ducharme, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 015117
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Asthma
Keywords: asthma; children; adolescent; education; medical review; asthma control; questionnaire; quality of life; emergency department visit; use of medication; adherence to treatment
MeSH Terms: conditions — Asthma; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asthma control awareness (Experimental): Multifaceted intervention to increase the patient awareness of the leve of asthma control
  Interventions: Procedure: asthma control awareness
- Usual care (Active Comparator): Usual care
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: asthma control awareness — Repeated assessments of the child's asthma control using the Asthma Quiz for Kidz, with recommendation for asthma education and medical visit
  Arms: Asthma control awareness
Procedure: Usual care — Recommendation for asthma education and/or follow-up at the physician's discretion
  Arms: Usual care

SUMMARY:
The objectives of this trials are to demonstrate, in children with poorly controlled asthma, that an intervention to increase the awareness and the impact of poor asthma control among parents and physicians of affected children and adolescents can reduce the rate of asthma emergency visits in the 12 months following the initiation of the intervention.

DETAILED DESCRIPTION:
In the philosophy of the "Programs to integrate information service and manage education(PRIISME)", the proposed randomised controlled trial will examine a novel approach based on education to trigger practice changes in community physicians and pharmacists as well as behavioural changes in parents of poorly controlled asthmatic children and in adolescents. Poorly controlled asthmatic children will be identified among those who present to the emergency department of the Montreal Children's Hospital for an acute asthma exacerbation. The novel approach hinges on alerting parents, physicians, pharmacists, and, for adolescents, the patients themselves, of the actual degree of asthma control and its impact on usual activities. The instrument used, the Asthma Quiz for Kidz, is a brief 5-item questionnaire based on the Canadian Asthma Consensus statement.

The tested intervention is comprised of (1) notifying by mail the treating physician of: the index emergency department or hospital admission, the results on the Asthma Quiz for Kidz in the month preceding the index exacerbation, the orientation of the patient to his/her local Asthma Education Centre (AEC), and the treatment protocol of the Canadian Asthma Consensus statement and providing a prescription pad containing the Asthma Impact Checklist; (2) referring the parents and child or adolescent to a personalised educational session with a highly trained asthma educator approved by the AEC, at a site identified closest to home or work; giving them a refrigerator magnet of the Asthma Quiz for Kidz; trimestrial mailing the 5-item Asthma Quiz for Kidz with a simple guide to interpret the degree of control, re-enforcing the message that control can be improved, and reminding them to consult their physician; (3) providing the identified AEC educator with a standard form, to be mailed to the treating physician and the co-ordinating centre, on which to record the results on the Asthma Quiz for Kidz, the interventions and recommendations made to the parents pertaining to environment, drug use, need to consult MD for an action plan; (4) providing pharmacists with a pad of the Asthma Quiz for Kidz to administer to identified patients at each request to refill asthma drugs.

The control intervention is the current usual care with referral of all hospitalised patients to the Montreal Children's Hospital (MCH) asthma educator (current attendance rate of 30%) and referral of non-hospitalised children to the MCH Asthma Centre, at the discretion of the emergency physicians.

The primary outcome is the rate of emergency department visits in the 12 months post-randomisation. Secondary outcomes include others measures of health care resources utilisation (hospital admission, physician's visits), measures of appropriateness of asthma drug use (refill rate of reliever drugs, ratio of inhaled preventer/reliever drugs, rate of rescue systemic steroids), and quality of life measures (for the school-aged child and the caregiver).

If proven effective in reducing asthma morbidity, the current strategy may be implemented at relatively low cost, relative to the savings in health care expenditures for poorly controlled asthmatic children. This intervention could then be tested in other populations and settings.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 17 years of
* acute asthma requiring emergency room visit or hospital admission
* understanding of French or English

Exclusion Criteria:

1. the index exacerbation is the first episode of wheezing in the previous year,
2. there is co-existence of other chronic pulmonary (such as Bronchopulmonary dysplasia (BPD), cystic fibrosis (CF)), renal or cardiac diseases;

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 298 (Actual)
Dates: Start 2002-08; Primary Completion 2007-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
rate of emergency department (ED) visits per person-month of observation, derived from Quebec provincial database (RAMQ) data. | 1 year
  rate of ED visit derived from provincial administrative databases

SECONDARY OUTCOMES:
Usage of asthma medication (refill rate of reliever drugs, ratio of reliever/preventer drugs; rate of rescue systemic steroids) as assessed from pharmacy records and RAMQ data | 1 year after randomisation
  use of medication based on data claims from provincial administrative databases
Quality of life of the child and caregivers using Juniper's instruments | 1 year after randomisation
  QOL measured on the Juniper questionnaires, measured at 12 months.
Change in asthma control between baseline and 12 months | 1 year after randomisation
  Change in Asthma Quiz for Kidz score between baseline and 12 months
Health care resources utilisation for asthma care (hospitalisation for asthma, hospitalisation for any cause, ratio of clinic to emergency department, as reflection of the ratio of preventive over curative care). | 1 year after randomisation
  Use of healthcare services based on data claims from provincial administrative databases

CONTACTS AND LOCATIONS:
Overall Officials: Francine M. Ducharme, MD, MSc, Principal Investigator — CHUS-Ste Justine Hospital
Locations (1):
- Ste-Justine Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided